CLINICAL TRIAL: NCT04851002
Title: Analysing the Effects of Advanced-platelet Rich Fibrin and Concentrated Growth Factor on Implant Osseointegration With Respect to the Levels of TNF-α, RANKL, and OPG in Peri-implant Crevicular Fluid: a Split-mouth Design Study
Brief Title: Effects of Different Centrifuged Platelet Concentrates on Bone Remodelling Around Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammet Atilgan (Other)
Collaborators: Mustafa Kemal University (Other)
Responsible Party: Sponsor-Investigator, Muhammet Atilgan, Researcher, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20.U.002
Record Dates: First submitted 2021-04-05; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Edentulous Jaw; Bone Loss, Alveolar; Resorption, Bone
Keywords: Concentrated Growth Factor; Advanced Platelet Rich Fibrin; Inflammatory Cytokines; Implant Osseointegration; Peri-implant Crevicular Fluid
MeSH Terms: conditions — Jaw, Edentulous; Alveolar Bone Loss; Bone Resorption | interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: This is a split-mouth design study. Accordingly, our study was conducted on 40 patients, including 20 patients in the CGF(Concentrated Growth Factor) study group and 20 patients in the A-PRF(Advanced Platelet Rich Fibrin) study group. While the implant combined with any regenerative material (CGF or A-PRF) was applied to the test site randomly assigned in the mouth, dental implants were placed according to traditional methods without applying any additional material to the contralateral site. Implants were placed symmetrically in the region of incisors, premolars or molar teeth in the mandible.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group in which the patients were included was determined by pulling the closed envelope just before the surgery. Test side was determined by tossing a coin after the implant cavities were prepared but before the implants were placed. The examiners who carried out the measurements and analyzes were unaware of the study and the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CGF TEST GROUP (Experimental): Concentrated growth factor liquid applied into the implant cavity. Also CGF membrane covered the implant and the socket. That is the only difference between CGF control group and CGF test group
  Interventions: Procedure: Application of concentrated growth factor with dental implants
- A-PRF TEST GROUP (Experimental): Advanced Platelet Rich Fibrin liquid applied into the implant cavity. Also A-PRF membrane covered the implant and the socket. That is the only difference between A-PRF control group and A-PRF test group
  Interventions: Procedure: Application of advanced platelet rich fibrin with dental implants
- CGF CONTROL GROUP (Experimental): Dental implant applications were made with traditional methods.
  Interventions: Procedure: Control side of concentrated growth factor study group
- A-PRF CONTROL GROUP (Experimental): Dental implant applications were made with traditional methods.
  Interventions: Procedure: Control side of advanced platelet rich fibrin study group

INTERVENTIONS:
Procedure: Application of concentrated growth factor with dental implants — Concentrated growth factor(CGF) liquid applied to the implant cavity also CGF membrane covered socket and implant
  Arms: CGF TEST GROUP
Procedure: Application of advanced platelet rich fibrin with dental implants — Advanced platelet rich fibrin (A-PRF) liquid applied to the implant cavity also A-PRF membrane covered socket and implant
  Arms: A-PRF TEST GROUP
Procedure: Control side of concentrated growth factor study group — Traditional implant methods applied
  Arms: CGF CONTROL GROUP
Procedure: Control side of advanced platelet rich fibrin study group — Traditional implant methods applied
  Arms: A-PRF CONTROL GROUP

SUMMARY:
Platelet concentrates obtained from blood have been used as regenerative biomaterials in periodontal surgery. Along with the migration and proliferation of osteogenic cells, platelets accelerate bone regeneration by increasing the formation of blood vessels and inducing inflammatory reactions. Experimental studies revealed that growth factors released from platelets enhance osteoblastic differentiation on the implant surface, and enlarge the contact surface of the bone and implant. Platelet-rich fibrin (PRF), a platelet concentrate, was introduced by Choukroun in 2001, and it contains a significant amount of cytokines. Advanced-platelet rich fibrin (A-PRF), discovered in 2014, is a PRF derivative with a denser leukocyte concentration and a softer consistency. Concentrated growth factor (CGF), another platelet derivative, differs from A-PRF since it contains many concentrated growth factors trapped in a more rigid fibrin structure. It was reported that both A-PRF and CGF, obtained with variable centrifuge speeds, accelerated the proliferation and differentiation of bone cells.

Stimulated osteoblasts and osteocytes initiate the remodelling process by producing macrophage colony-stimulating factor and receptor activator of nuclear factor-kappa B ligand (RANKL).Previous studies reported that TNF-α initiated bone resorption independently of RANKL.Osteoprotegerin (OPG) is a soluble cytokine receptor of the TNF family and is produced by osteoblasts, fibroblasts, and a number of host cells. OPG binds to RANKL and prevents the RANKL-RANK interaction Therefore, it inhibits osteoclastic activity. The RANKL/OPG ratio is used as an indicator for estimating bone remodelling, osteoclastic activity, or osteogenesis.

The interactions among cytokines, growth factors, chemokines, and chemical mediators during blood clot formation result in a complex signalling process. High concentrations of cytokines and growth factors in the wound promote the migration of macrophages, neutrophils, and lymphocytes. Therefore, it was reported that the cytokines released from the fibrin matrix might affect those signaling pathways. In this study, investigators hypothesised that the application of CGF or A-PRF in dental implantation would contribute to inflammation, proliferation and the remodeling process. Therefore, the aim of this study was to investigate the effects of CGF and A-PRF on the osseointegration of dental implants in clinical, radiographic, and biochemical aspects.

DETAILED DESCRIPTION:
This study was conducted in Periodontology clinics. The study protocol was approved by the Hatay Mustafa Kemal University Human Ethics Committee before the initiation of the study (approval number:). The patients who met the inclusion criteria and who volunteered to participate in the study were given detailed information about the study and provided informed consent before the procedure.

Patient selection:

The inclusion criteria of the individuals found to be healthy from their medical histories and who had received clinical examination and had radiological imaging were as follows:

* Above 18 years of age
* Symmetrical edentulous areas in the mandible
* Sufficient bone width and height permitting ideal dental implant placement
* Individuals who do not smoke
* At least 2 mm of keratinized gingiva width and 3 mm soft tissue thickness at the implant site

Individuals meeting any of the criteria listed below were excluded from the study:

* Patients with systemic disorders, including diabetes mellitus, metabolic bone disease, rheumatoid arthritis, mucocutaneous disorders, immunological disorders, hepatitis, or HIV
* Individuals who were on antibiotics, anti-inflammatory agents, corticosteroids, immunosuppressants, anticoagulants, or hormonal contraceptives for any reason, at least 6 months prior to the procedure, and those who were on bisphosphonates at that time or previously.
* Individuals with any pathology or defects at the implant site.
* History augmentation at the implant site.
* Individuals with severe periodontal disease and poor oral hygiene.
* Severe caries or endodontic lesions in teeth adjacent to the implant.
* Those who use intraoral orthodontic or prosthetic appliances that make plaque control difficult.
* Pregnant and lactating individuals. Randomization and Blinding Both the study groups and the surgical site were determined by drawing a closed envelope immediately before surgery. Clinical and radiological records of the study were obtained by an experienced periodontist who was unaware of the allocation

Surgical Procedure

Infiltrative anaesthesia was provided with an anaesthetic solution containing 1:100,000 epinephrine. A mid-crestal incision was made using a 15c scalpel, and a full-thickness flap was elevated. The drilling procedure was performed (600 rpm and 25 Ncm) according to the implant diameter and the need for an edentulous area in the mandible. A countersink drill was used for all implants to minimise the crestal bone stress. In case of the presence of a natural tooth adjacent to the implant site, a distance of at least 1.5 mm between the tooth and the implant cavity was left, and the presence of at least 1 mm bone plates in the buccal and lingual sides of the implant. CGF or A-PRF autologous obtained from centrifuged blood was placed in a PRF box. In this way, the liquid rich in growth factor and platelets leaking from the fibrin network was allowed to flow into the box. The liquid was collected with a syringe and applied over the implant surface until no dry area was left. In addition, the implant site was filled with this liquid, and 0.5 mm subcrestal placement of the implant was provided at 40 rpm and 25 Ncm torque. The membrane obtained from the CGF or A-PRF was placed over the implant, enough to cover the crestal bone, and a healing cap was placed. Implant placement without CGF or A-PRF was performed on the opposite side of the jaw in the control group. The stability of the implant was determined using resonance frequency analysis. The surgical site was sutured using a 5/0 silk. All patients were advised not to take any medications, unless necessary. The sutures were removed at the 10 days after surgery. All surgeries were performed by a physician with five years of experience Preparation Procedure of CGF and A-PRF Before starting the implant surgery, 9 mL of blood was withdrawn from the cubital vein of the patient's forearm, transferred into a tube without anticoagulant, and centrifuged. CGF was obtained using an automatically adjusted centrifuge device, fired at alternating and controlled speeds (2 min at 2700 rpm, 4 min at 2400 rpm, 4 min at 2700 rpm, and 3 min at 3000 rpm) (MEDIFUGE, Silfradentsrl, S. Sofia, Italy). In the A-PRF group, blood was centrifuged at 1400 rpm for 14 min (Duo Centrifuge Process for PRF, France). Centrifugation resulted in three layers in the tube: a red blood cell layer at the bottom, a platelet-poor serum layer at the top, and a fibrin gel layer containing growth factors and platelets in the middle. The serum in the upper layer was removed with a sterile syringe, and the fibrin layer was removed from the tube using a clamp. The red blood cells in the lower layer were removed from the fibrin structure using a scissors.

Clinical Measurements and Resonance Frequency Analysis Four sites of each healing cap, mesial, distal, buccal, and lingual surfaces, were analysed for plaque index (PI), gingival index (GI), pocket depth (PD), and gingival bleeding index (GBI). All clinical measurements were repeated at 2, 4, and 12 weeks after the procedure. Resonance frequency analysis was performed intraoperatively and postoperatively at the fourth and twelfth month.

Measurement of Marginal Bone Levels:

Calibrated panoramic radiographs obtained on the day of surgery and 3 months after were used to determine the marginal bone level. The implant-fixture platform was considered as the threshold for measuring changes in the marginal bone level. When the marginal bone around the dental implant decreased below the platform, two horizontal lines were drawn on the radiograph: the first plane was located on the platform of the implant fixture, and the second was on the alveolar crest or at the bottom of the bone defect. The average of the marginal bone loss was obtained by measuring the distance between the two points left by the lines drawn from the mesial and distal surfaces of the cylindrical part of the implant on the horizontal lines. All radiological measurements were performed by two examiners experienced in their fields.

Collection of Peri-implant Crevicular Fluid (PICF):

First, the implant site was isolated from saliva and dried with air. An absorbent filter paper strip was placed 1 mm into the pocket in the mesial and distal surfaces of the healing cap, and was left there for 30 s to allow absorption of a sufficient amount of peri-implant crevicular fluid. The volume of the fluid was measured using a calibrated electronic device (Periotron 8010, Oraflow, Amityville, NY, USA). Paper strips contaminated with blood or plaque were excluded from the study. The paper strips were transferred into an empty Eppendorf tube covered with paraffin wax and stored at 80 °C until analysis.

Biochemical Analysis:

Initially, fresh phosphate buffered saline (PBS) was prepared saline (pH: 7.00 137 mM NaCl, 10 mM Na2HPO4, and 2.7 mM KCl]. PBS of 300 µL) was added to each Eppendorf tube with two paper strips inside, left at room temperature for 30 min, and then centrifuged at 12,000 × g at 4°C for 15 min. Following centrifugation, the strips in the Eppendorf tube were removed, and the supernatant obtained was used for ELISA. Tumour necrosis factor alpha (TNF-α) (Boster), sRANKL (Soluble Receptor Activator of Nuclear Factor-Kb Ligand) (Elabscience) and Osteoprotegerin (OPG) (Boster) levels were measured by ELISA at 450 nm wavelength using commercial kits and Thermo Fisher Scientific Multiscan Go- Finland ELISA Reader. All analyses were performed in accordance with the manufacturer's instructions.

Statistical Analysis:

The data were analysed at 95% confidence using the SPSS 21 software. Continuous variables were expressed as mean, standard deviation, median, minimum, and maximum. Categorical variables are expressed as frequencies and percentages. The normality of the distribution of the data was analysed using the Shapiro-Wilk test, and Mann Whitney U and Student t tests were used to compare independent groups. The Wilcoxon signed rank test and Friedman test were used to compare dependent variables. The comparisons of two measurement points were analysed using the Wilcoxon test with Bonferroni correction (p <0.016) if a significant difference was determined using the Friedman test. The p value was determined as 0.05, for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Symmetrical edentulous areas in the mandible
* Sufficient bone width and height permitting ideal dental implant placement
* Individuals who do not smoke
* At least 2 mm of keratinized gingiva width and 3 mm soft tissue thickness at the implant site

Exclusion Criteria:

* Patients with systemic disorders, including diabetes mellitus, metabolic bone disease, rheumatoid arthritis, mucocutaneous disorders, immunological disorders, hepatitis, or HIV
* Individuals who were on antibiotics, anti-inflammatory agents, corticosteroids, immunosuppressants, anticoagulants, or hormonal contraceptives for any reason, at least 6 months prior to the procedure, and those who were on bisphosphonates at that time or previously.
* Individuals with any pathology or defects at the implant site.
* History augmentation at the implant site.
* Individuals with severe periodontal disease and poor oral hygiene.
* Severe caries or endodontic lesions in teeth adjacent to the implant.
* Those who use intraoral orthodontic or prosthetic appliances that make plaque control difficult.
* Pregnant and lactating individuals.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Loss | Third month
  Marginal bone loss measured around dental implants from mesial and distal surfaces on panoramic radiography obtained at the third month of the study.
Resonance Frequency Analysis-I | Immediately after surgery
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
Resonance Frequency Analysis-II | Fourth week
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
Resonance Frequency Analysis-III | Third month
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
TNF-alpha-I | Second week
  TNF-alpha isolated from peri-implanter crevicular fluid. The level of TNF-alpha has been analyzed by ELISA, and its level was determined as pg/dL
TNF-alpha-II | Fourth week
  TNF-alpha isolated from peri-implanter crevicular fluid. The level of TNF-alpha has been analyzed by ELISA, and its level was determined as pg/dL
TNF-alpha-III | Third month
  TNF-alpha isolated from peri-implanter crevicular fluid. The level of TNF-alpha has been analyzed by ELISA, and its level was determined as pg/dL
RANKL-I | Second week
  RANKL isolated from peri-implanter crevicular fluid. The level of RANKL has been analyzed by ELISA, and its level was determined as pg/dL
RANKL-II | Fourth week
  RANKL isolated from peri-implanter crevicular fluid. The level of RANKL has been analyzed by ELISA, and its level was determined as pg/dL
RANKL-III | Third month
  RANKL isolated from peri-implanter crevicular fluid. The level of RANKL has been analyzed by ELISA, and its level was determined as pg/dL
OPG-I | Second week
  OPG isolated from peri-implanter crevicular fluid. The level of OPG has been analyzed by ELISA, and its level was determined as pg/dL
OPG-II | Fourth week
  OPG isolated from peri-implanter crevicular fluid. The level of OPG has been analyzed by ELISA, and its level was determined as pg/dL
OPG-III | Third month
  OPG isolated from peri-implanter crevicular fluid. The level of OPG has been analyzed by ELISA, and its level was determined as pg/dL
RANKL/OPG ratio-I | Second week
  RANKL/OPG ratio is important for analysing bone remodeling and resorption process. RANKL/OPG ratio is obtained by dividing the RANKL level to the OPG level.
RANKL/OPG ratio-II | Fourth week
  RANKL/OPG ratio is important for analysing bone remodeling and resorption process. RANKL/OPG ratio is obtained by dividing the RANKL level to the OPG level.
RANKL/OPG ratio-III | Third month
  RANKL/OPG ratio is important for analysing bone remodeling and resorption process. RANKL/OPG ratio is obtained by dividing the RANKL level to the OPG level.

SECONDARY OUTCOMES:
Plaque Index-I | Second week
  The plaque index assesses the amount of around dental implant visible plaque amount on the four surfaces of an implant including mesial, distal, buccal and lingual.
Plaque Index-II | Fourth week
  The plaque index assesses the amount of around dental implant visible plaque amount on the four surfaces of an implant including mesial, distal, buccal and lingual.
Plaque Index-III | Third month
  The plaque index assesses the amount of around dental implant visible plaque amount on the four surfaces of an implant including mesial, distal, buccal and lingual.
Gingival Index-I | Second week
  This measurement is based on the presence or absence of bleeding on gentle probing. Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous. The four surfaces of the implant are assessed in the index system
Gingival Index-II | Fourth week
  This measurement is based on the presence or absence of bleeding on gentle probing. Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous. The four surfaces of the implant are assessed in the index system
Gingival Index-IIII | Third month
  This measurement is based on the presence or absence of bleeding on gentle probing. Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous. The four surfaces of the implant are assessed in the index system
Probing Depth-I | Second week
  A periodontal probe is used to measure the depths of gingival sulcus from six areas of each implant (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual), and the readings are recorded onto a chart
Probing Depth-II | Fourth week
  A periodontal probe is used to measure the depths of gingival sulcus from six areas of each implant (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual), and the readings are recorded onto a chart
Probing Depth-III | Third month
  A periodontal probe is used to measure the depths of gingival sulcus from six areas of each implant (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual), and the readings are recorded onto a chart
Gingival Bleeding Index-I | Second week
  Traditionally, bleeding on probing has been used to diagnose the presence of periodontal diseases, and it is a reliable indicator of gingival inflammation, especially when used in conjunction with other factors. After probing the gingival sulcus, the presence of bleeding is assessed dichotomously. If the bleeding occurs after probing (+), or (-).
Gingival Bleeding Index-II | Fourth week
  Traditionally, bleeding on probing has been used to diagnose the presence of periodontal diseases, and it is a reliable indicator of gingival inflammation, especially when used in conjunction with other factors. After probing the gingival sulcus, the presence of bleeding is assessed dichotomously. If the bleeding occurs after probing (+), or (-).
Gingival Bleeding Index-III | Third month
  Traditionally, bleeding on probing has been used to diagnose the presence of periodontal diseases, and it is a reliable indicator of gingival inflammation, especially when used in conjunction with other factors. After probing the gingival sulcus, the presence of bleeding is assessed dichotomously. If the bleeding occurs after probing (+), or (-).

CONTACTS AND LOCATIONS:
Overall Officials: Osman Fatih ARPAG, PhD, Study Director — Mustafa Kemal University
Locations (1):
- Mustafa Kemal University, Hatay, Turkey (Türkiye)